CLINICAL TRIAL: NCT06459024
Title: Master Framework For Relapse or Refractory Acute Myeloid Leukemia- IMPACT STREAM - A Prospective Observational Study of Treatment Outcomes
Brief Title: Master Framework For Relapse or Refractory Acute Myeloid Leukemia
Acronym: IMPACT STREAM
Status: Recruiting | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Hospital Vall d'Hebron (Other); Cyprus Institute of Neurology and Genetics (Other); European LeukemiaNet (Network); Fundacion Para La Investigacion Hospital La Fe (Other); Ostedusche Hematology and Oncology Study Group (Unknown); Ospedale Pediatrico Bambin Gesù (Other); Czech Lymphoma Study Group (Other); Charite University, Berlin, Germany (Other); Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other); University of Bologna (Other); Hannover Medical School (Other); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Toscana Life Sciences Sviluppo s.r.l. (Industry); Lithuanian University of Health Sciences (Other); Gruppo Italiano Malattie EMatologiche dell'Adulto (Other); Time.Lex (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRST204.08
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
Keywords: Relapsed; Refractory; Acute Myeloid Leukemia; Framework
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with relapsed or refractory acute myeloid leukemia: All patients with relapsed or refractory acute myeloid leukemia
  Interventions: Other: Registration into the STREAM platform

INTERVENTIONS:
Other: Registration into the STREAM platform — All patients fulfilling eligibility criteria will be registered into the STREAM platform. Baseline and follow up information will be recorded for each patient enrolled. Each patient will be followed up according to normal clinical practice up to 4 years.

SUMMARY:
This is an observational (non-interventional), prospective, cohort study that will collects data from patients diagnosed with relapsed or refractory acute myeloid leukemia afferent to the participanting clinical sites

DETAILED DESCRIPTION:
Treatment outcome for acute myeloid leukemia (AML) has improved over the last few decades. With intensive multidrug induction regimens, a complete remission is expected. Despite such advances, therapy resistance or relapse remains the main causes of death in adult patients and in children. Relapsed or refractory (R/R) AML is a hard-to-treat disease, with a 5-year overall survival (OS) estimate below 20% in adults and 30%-35% in children, and no standard of care exists. HSCT (allogeneic hematopoietic stem cell transplantation) remains the only curative strategy for R/R AML patients, including pediatric and elderly ones. Some new personalized therapies have recently been integrated into the treatment options of R/R AML. However, there is a need to collect consistent data on the efficacy of these new strategies in real-world settings. Lack of data from clinical trials can be a barrier in most countries, limiting patient accessibility to some very effective drugs. The STREAM study is part of the Horizon Europe Mission Cancer 2022 IMPACT-AML project, that proposes to create an inclusive master framework for relapsed or refractory acute myeloid leukemia. In STREAM we will collect data and monitor outcomes of patients with R/R AML across Europe. In close collaboration with the European Reference Network on Rare Hematological Diseases (ERN-EuroBloodNet, GA101157011), STREAM is developed under ERN-EuroBloodNet central registry, the European Rare Blood Disorders Platform (ENROL), incorporating EU standards for interoperability and the GPDR-compliant SPIDER pseudonymization tool offered by the EU-RD Platform in the context of rare disease registries will be implemented, to allow cross-hospital and cross-country participation. The STREAM study will allow to collect high-quality data from patients at any stage of the disease, for any cancer subtype, in any age group, including pediatric and elderly population, unfit patients, patients with rare mutations, patients with high-impact end-organ damage, patients from rural regions, post-transplant relapse. Data collected in STREAM will foster the production of novel knowledge on rare populations in a pragmatic setting and will form the basis for building international trials to be conducted worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML diagnosis according to WHO2022 or ICC2022
* Treatment failure (i.e. relapse, refractory or progression, including MRD) according to ELN2022 criteria
* Participant or his/her legal representative is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Patients included in clinical trials may be enrolled except where otherwise specified in the experimental protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsed or refractory acute myeloid leukemia
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to determine the overall survival of R/R AML patients | 8 years
  Overall survival is defined as the time from R/R diagnosis to death due to any cause.

SECONDARY OUTCOMES:
Remission rate | 8 years
  Response is defined according to ELN 2022 criteria. Rates of CR, CRi, CRh and overall response (CR+CRi+CRh) as best response will be considered
Event-free survival | 8 years
  Event-free survival is defined as the time from R/R diagnosis to rescue treatment failure (according to ELN 2022 definitions), relapse or death due to any cause, whichever occurs first.
Relapse free survival | 8 years
  Relapse-free survival is defined for patients achieving a response to rescue treatment as the time from response onset to relapse or death due to any cause, whichever occurs first.
Transplant rate | 8 years
  Proportion of patients undergoing transplantation
Describe the methods for diagnosis and the treatment options offered to the patients affected by R/R AML | 8 years
  type and frequency of diagnostic procedures used and treatments prescribed
Association between baseline clinical, molecular and biological parameters and clinical outcomes | 8 years
  Rates of CR, CRi, CRh and overall response (CR+CRi+CRh) in specific sub-populations bearing common molecular features
To characterize potential populations that could be target for future studies/clinical trials | 8 years
  descriptive statistics (mean, median, frequency, range) of subpopulations characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Prof, Study Chair — University of Bologna
Locations (38):
- Germany (4):
  - University Hospital Aachen, Aachen
  - University Hospital Greifswald, Greifswald
  - University Hospital Halle, Halle
  - University Hospital of Rostock, Rostock
- Italy (30):
  - Policlinico Sant'Orsola-Malpighi, Bologna, BO
  - Ospedale "A. Perrino", Brindisi, BR
  - ASST Spedali Civili, Brescia, BS
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Ospedale Valduce, Como, CO
  - ASST Cremona, Cremona, CR
  - AOU Universitaria Arcispedale Sant'Anna, Ferrara, FE
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo, PA
  - Presidio Ospedaliero "Santo Spirito", Pescara, PE
  - Ospedale Santa Maria della Misericordia, Perugia, PG
  - Ospedale Santa Maria delle Croci, Ravenna, RA
  - Fondazione Policlinico Tor Vergata, Roma, RM
  - Policlinico Umberto I, Roma, RM
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma, RM
  - Ospedale Sant'Andrea, Roma, RM
  - Ospedale infermi di Rimini, Rimini, RN
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno, SA
  - AOU Città della Salute e della Scienza di Torino, Torino, TO
  - AO Ordine Mauriziano, Torino, TO
  - IOV Istituto Oncologico Veneto, Castelfranco Veneto, TV
  - ASST Valle Olona, Busto Arsizio, VA
  - AOU Careggi, Florence
  - IRST Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli
  - AOU Maggiore della Carità, Novara
  - Azienda Ospedale-Università Padova, Padua
  - Ospedale San Bortolo, Vicenza
- The Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Lithuania
- University Clinical Center in Gdańsk, Gdansk, Poland
- Fundeni Clinical Institute, Bucharest, Romania
- University Hospital La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No